CLINICAL TRIAL: NCT05825183
Title: Study of Product of Conception Derived From Ultrasound-guided Manual Vacuum Aspiration
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2023.095
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Genetic Anticipation; Immunological Abnormalities
MeSH Terms: conditions — Anticipation, Genetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ultrasound-guided manual vaccum — For managing with miscarriage or termination of pregnancy (TOP) in first trimester loss, ultrasound-guided manual vacuum aspiration (USG-MVA) is one of the treatment options.
  The USG-MVA device works by aspirating the uterine content via the cannula into the syringe. Furthermore, product of conception derived from USG-MVA can be sent for karyotyping analysis.
  POCs obtained from MVA procedure were rinsed in normal saline thoroughly in the kidney basin to minimize maternal blood. Chorionic villi were considered as a proxy of fetal genetics, appeared to be yellowish in color and tree-projection-like in appearance, floating on the surface of the waterline. Decidua are originated from the mother, appeared substantive in structure and sank in the basin. The two different types of tissues are separated from each other for different testing.

SUMMARY:
Early pregnancy loss is very common, approximately one in four women will experience a miscarriage in their lifetime. The etiology of pregnancy loss remains largely unknown, although genetic, anatomical, endocrinological and immunological abnormalities have been implicated.

It is known that embryonic/fetal chromosomal aberrations contributed to approximately 50% of early pregnancy loss, among which 60-70% were aneuploidies, largely can be detected by the current gold standard karyotyping approach recommended by various international societies. However, the drawbacks of conventional karyotyping include the risk of culture failure, maternal cell contamination (MCC), limited detection resolution (5-10 Mb), and differential growth of specific cell lineages which could hinder the diagnosis of genetic abnormalities, particularly mosaicisms. Additional genetic factors beyond the resolution of karyotyping are not well studied.

DETAILED DESCRIPTION:
Early pregnancy loss is very common, approximately one in four women will experience a miscarriage in their lifetime. The etiology of pregnancy loss remains largely unknown, although genetic, anatomical, endocrinological and immunological abnormalities have been implicated.

It is known that embryonic/fetal chromosomal aberrations contributed to approximately 50% of early pregnancy loss, among which 60-70% were aneuploidies, largely can be detected by the current gold standard karyotyping approach recommended by various international societies. However, the drawbacks of conventional karyotyping include the risk of culture failure, maternal cell contamination (MCC), limited detection resolution (5-10 Mb), and differential growth of specific cell lineages which could hinder the diagnosis of genetic abnormalities, particularly mosaicisms. Additional genetic factors beyond the resolution of karyotyping are not well studied.

Next-generation sequencing (NGS) has brought genetic testing to new frontiers, expanding the scope of detectable genomic variants. Moreover, its significant reduction in costs over the years has facilitated the implementation of genetic diagnostic testing. Our customized shallow read-depth genome sequencing analytical pipeline, namely low-pass genome sequencing (GS), enables efficient and cost-effective detection of genome-wide copy-number variants (CNVs, >50 kb) and low-level chromosomal mosaicisms (as low as 10%). Furthermore, the roles of cryptic structural rearrangements, absence of heterozygosity (AOH), and single-nucleotide variant (SNV) were less understood in current studies.

Various versions of sequencing platforms targeting at different variants were already established and validated in the Prenatal Genetic Diagnostic Laboratory, The Chinese University of Hong Kong, including FetalSeq, ChromoSeq, and 30xWGS.

Human endometrial and decidual tissues, containing a myriad of immune and inflammatory populations, are immunologically dynamic. In the early proliferative phase of the menstrual cycle, T-cells are the most abundant leukocyte population in the endometrium, but they decrease to 20% of all stromal leukocytes during early pregnancy. Macrophages are also present in endometrial tissues during all phases of the menstrual cycle, but are most abundant in late secretory endometrium and in decidual tissues during early pregnancy. The most abundant population (70%) of stromal leukocytes observed in late secretory endometrium and in the decidua during early normal pregnancy are large granular lymphocytes (LGL) bearing the unique phenotype: CD56++, CD16-, CD57-, CD2±, CD38±, CD3-, CD4-, CD8-. Increased mean numbers of CD56+ cells have been reported in secretory endometrium of women with recurrent miscarriages.

The hypothesis that the balance between T-cell subsets (i.e. CD4+ and CD8+ cells) plays a role in maintaining successful pregnancy is controversial. Some studies have reported no difference between the proportions of T-cell subsets in either secretory endometrium or first trimester decidua from women with a history of recurrent pregnancy loss compared with normal controls; while others have described a shift towards a higher ratio of CD8+ T-cells in endometrial biopsies from women with a history of recurrent pregnancy loss.

The activation status of T-cell populations may provide another indicator of cellular immunity potentially involved in pregnancy loss. The IL-2 receptor has been reported to be absent on T-cells in normal first trimester decidual tissues using immunohistochemical techniques; however, using flow cytometry, CD3+CD25+ activated T-cells have been identified in decidual tissue. CD69 is another early activation marker expressed on the surface of T-cells. A proportion of T-cells constitutively expresses this marker throughout the menstrual cycle and in normal early pregnancy.

Approximately 60% of spontaneous abortions are attributable to numerically abnormal chromosomes in the developing conceptus, yet limited data to date addressing immunological phenomena in the decidua of miscarried women has compared their data relative to well-defined chromosomal abnormalities belonging to conceptuses. This is important since the chromosome abnormality trisomy 16, which occurs in 26% of all spontaneous abortions, is incompatible with life and would thus be an undisputed cause of spontaneous abortion. Therefore, the purpose of our study was to determine whether decidual leukocyte subpopulations and their associated activation markers were different between women having miscarriage of either a trisomy 16 conceptus (47XY+16 or 47XX+16) compared with a chromosomally normal male conceptus (46XY) and compared with gestationally age-matched decidual tissues. Samples from presumably normal female conceptuses (46XX) were not chosen for study because of the inability to accurately differentiate from possible maternal cell contamination.

For managing with miscarriage or termination of pregnancy (TOP) in first trimester loss, ultrasound-guided manual vacuum aspiration (USG-MVA) is one of the treatment options. USG-MVA for the treatment of early pregnancy loss has been used for many decades. It had been reported that USG-MVA is safer, more cost-effective, and is associated with shorter hospitalization time and cost than surgical evacuation under general anesthesia . USG-MVA is a surgical technique of suction curettage. It is performed by using a hand held vacuum source (a syringe with barrel and plunger) attached to a uterine cannula. The USG-MVA device works by aspirating the uterine content via the cannula into the syringe. Furthermore, product of conception derived from USG-MVA can be sent for karyotyping analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years old or above
2. Women with miscarriage or TOP who are suitable candidates for MVA

   * first trimester miscarriage or TOP
   * No fetal heart beat or TOP in those with CRL 25mm
   * incomplete miscarriage or TOP with POG <5cm
   * hemodynamically stable,
   * tolerates well with speculum examination

Exclusion Criteria:

1. Women who are not feasible for the MVA procedure

   * cervical stenosis
   * fibroid uterus >12 weeks in size
   * known uterine malformation
   * bleeding disorder
   * clinically sepsis
   * inability to tolerate pelvic examination
2. History of psychological/ psychiatric problem
3. Patient refusal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Study Population: Women undergoing ultrasound-guided manual vacuum aspiration (USG-MVA) will be recruited at Obstetrics and Gynaecology in The Prince of Wales Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Histopathologic diagnosis of chorionic villi | 31 May 2028
  Detecting site-to-site heterogeneity and detecting cryptic structural rearrangements, absence of heterozygoisity (AOH), and single-nucleotide variant (SNV).
Immunohistochemistry staining | 31 May 2028
  immunoassay of maternal decidua

CONTACTS AND LOCATIONS:
Overall Officials: Pui Wah Jacqueline Chung, Principal Investigator — Prince of Wales Hospital
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WARBURTON D, FRASER FC. SPONTANEOUS ABORTION RISKS IN MAN: DATA FROM REPRODUCTIVE HISTORIES COLLECTED IN A MEDICAL GENETICS UNIT. Am J Hum Genet. 1964 Mar;16(1):1-25. No abstract available. PMID 14131871
- [Background] Klentzeris LD, Bulmer JN, Warren MA, Morrison L, Li TC, Cooke ID. Lymphoid tissue in the endometrium of women with unexplained infertility: morphometric and immunohistochemical aspects. Hum Reprod. 1994 Apr;9(4):646-52. doi: 10.1093/oxfordjournals.humrep.a138564. PMID 7519197
- [Background] Bulmer JN, Morrison L, Longfellow M, Ritson A, Pace D. Granulated lymphocytes in human endometrium: histochemical and immunohistochemical studies. Hum Reprod. 1991 Jul;6(6):791-8. doi: 10.1093/oxfordjournals.humrep.a137430. PMID 1757516
- [Background] Bulmer JN, Sunderland CA. Immunohistological characterization of lymphoid cell populations in the early human placental bed. Immunology. 1984 Jun;52(2):349-57. PMID 6376338
- [Background] Starkey PM, Sargent IL, Redman CW. Cell populations in human early pregnancy decidua: characterization and isolation of large granular lymphocytes by flow cytometry. Immunology. 1988 Sep;65(1):129-34. PMID 3181993
- [Background] Hill JA, Melling GC, Johnson PM. Immunohistochemical studies of human uteroplacental tissues from first-trimester spontaneous abortion. Am J Obstet Gynecol. 1995 Jul;173(1):90-6. doi: 10.1016/0002-9378(95)90175-2. PMID 7631733